CLINICAL TRIAL: NCT04488705
Title: A First in Human, Randomised, Double Blind, Placebo-controlled, Three-part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses (SAD & MAD) of Inhaled ETD002 in Healthy Male and Female Subjects
Brief Title: A First in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Inhaled ETD002 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enterprise Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-TMEM-01; 2020-001080-92 (EudraCT Number)
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single ascending dose (Experimental)
  Interventions: Drug: ETD002 - single dose; Drug: Placebo - single dose
- Repeat dose - 7 days (Experimental)
  Interventions: Drug: ETD002 - 7 day repeat dose; Drug: Placebo - 7 day repeat dose
- Repeat dose - 14 days (Experimental)
  Interventions: Drug: ETD002 - 14 day repeat dose; Drug: Placebo - 14 day repeat dose
- Repeat dose - 7 days with SABA (Experimental)
  Interventions: Drug: ETD002 - 7 day repeat dose; Drug: Placebo - 7 day repeat dose; Drug: Salbutamol

INTERVENTIONS:
Drug: ETD002 - single dose — Single ascending doses of ETD002
  Arms: Single ascending dose
Drug: Placebo - single dose — Single doses of placebo
  Arms: Single ascending dose
Drug: ETD002 - 7 day repeat dose — Twice daily doses of ETD002 for 7 days
  Arms: Repeat dose - 7 days; Repeat dose - 7 days with SABA
Drug: Placebo - 7 day repeat dose — Twice daily doses of Placebo for 7 days
  Arms: Repeat dose - 7 days; Repeat dose - 7 days with SABA
Drug: ETD002 - 14 day repeat dose — Twice daily doses of ETD002 for 14 days
  Arms: Repeat dose - 14 days
Drug: Placebo - 14 day repeat dose — Twice daily doses of Placebo for 14 days
  Arms: Repeat dose - 14 days
Drug: Salbutamol — Twice daily doses of salbutamol for 3 days (Days 5, 6 & 7)
  Arms: Repeat dose - 7 days with SABA

SUMMARY:
This is a first in human study of ETD002 a new drug being developed for the treatment of cystic fibrosis.The study is a randomised, double-blind, placebo-controlled, interventional study to assess the safety and tolerability of ascending single and repeat doses of inhaled ETD002 in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males & females using suitable methods of contraception or females of non-childbearing potential
* Consent to study participation
* Body weight ≥ 50 kg and body mass index within the range 19 - 30 kg/m2
* Vital signs assessments within normal ranges
* Healthy as determined following physical examination at screening visit
* Spirometry readings (FEV1 and FVC) to be ≥ 80% of predicted value

Exclusion Criteria:

* Acute or chronic illness detected at screening visit
* Respiratory tract infection within 4 weeks of the screening visit
* Use of prescription or OTC medication within 14 days of the screening visit
* History of regular alcohol consumption over recommended limits within 6 months of the study, or history/evidence of alcohol or drug abuse
* Smoking or use of tobacco products within 6 months of screening
* Abnormal blood/urine laboratory screening test results
* Current, or history of, allergy that may be contraindicated

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting one or more treatment emergent adverse event (TEAE) | Baseline to Week 8
Number of participants who discontinue due to an adverse event (AE) | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for 12-lead ECG assessment at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for vital signs assessments at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for safety laboratory assessments at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for spirometry assessments at least once post dose | Baseline to Week 8

SECONDARY OUTCOMES:
Plasma concentrations of ETD002 | Day 1 pre-dose and at multiple time points (up to 14 days) post final dose
  Blood levels of ETD002 measured after dosing

CONTACTS AND LOCATIONS:
Overall Officials: David Morris, MD, Study Director — Enterprise Therapeutics
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Miller P, Repplinger D, Zhu R, Chen Y, Lewin-Koh N, Morris D, Russell P, She G, Singh N, White R, Wilkes D, Chen H, Galanter J. Randomized, phase I studies to evaluate the safety, tolerability, and pharmacokinetics of an inhaled, TMEM16A potentiator, GDC-6988, in healthy subjects. Ther Adv Respir Dis. 2025 Jan-Dec;19:17534666251393346. doi: 10.1177/17534666251393346. Epub 2025 Nov 29. PMID 41318901